CLINICAL TRIAL: NCT00664690
Title: Effect of Celecoxib on Transitional Pain After Outpatient Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-04-309; 10457
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Pain
Keywords: shoulder surgery; analgesia
MeSH Terms: conditions — Pain; Agnosia | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): celebrex
  Interventions: Drug: celebrex
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: celebrex — 400 mg celebrex given 1 hour preop and celebrex 200 mg BID postop
  Arms: 1
Drug: placebo — placebo given preop and BID postop
  Arms: 2

SUMMARY:
Sixty adults having shoulder and forearm surgery will receive either placebo or celebrex started preoperatively and continued for 3 days. Rescue medications required as well as pain scores will be assessed using a patient diary to evaluate the effect of celebrex in controlling transitional pain

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective ambulatory surgery of the shoulder
* ASA I - III
* Able to read English
* Male or female

Exclusion Criteria:

* Allergy to local anesthetic, Cox2, sulpha drug, acetaminophen or oxycodone
* Women who are pregnant or lactating and women of childbearing age and not following acceptable contraceptive precautions
* Any major medical or psychiatric problem
* Those with a known history of narcotic dependence, abuse or chronic narcotic intake
* Patients with known history of peptic ulcer or GI bleeding in the past, ulcers, congestive heart failure, angina or previous heart attack, coagulation problems, venous thrombosis, kidney or liver disease or strokes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
visual analogue score for pain | post-op period

SECONDARY OUTCOMES:
severity of nausea | post-op period

CONTACTS AND LOCATIONS:
Overall Officials: Ngozi Imasogie, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada